CLINICAL TRIAL: NCT02803424
Title: Comparison of Volume Controlled Ventilation and Autoflow-volume Controlled Ventilation in Robot-assisted Laparoscopic Radical Prostatectomy With Steep Trendelenburg Position and Pneumoperitoneum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2016-0311
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Robot-assisted Laparoscopic Radical Prostatectomy Undergoing General Anesthesia
Keywords: robot-assisted laparoscopic radical prostatectomy; Autoflow; trendelenburg position; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volume controlled ventilation (Experimental): During the steep trendelenburg position and pneumoperitoneum, volume controlled ventilation will be applied with 8ml/kg (ideal body weight) and inspiration:expiration ratio (I:E) = 1:2.
  Interventions: Other: Volume controlled ventilation
- Autoflow-volume controlled ventilation (Active Comparator): During the steep trendelenburg position and pneumoperitoneum, Autoflow-volume controlled ventilation will be applied with 8ml/kg (ideal body weight) and inspiration:expiration ratio (I:E) = 1:2.
  Interventions: Other: Autoflow-volume controlled ventilation

INTERVENTIONS:
Other: Volume controlled ventilation — During anesthesia and surgical procedure, volume-controlled ventilation will be applied with an inspiration:expiration ratio of 1:2 and a tidal volume of 8 mL per ideal body weight (kg) without ventilatory mode change.
  Other Names: VCV
  Arms: Volume controlled ventilation
Other: Autoflow-volume controlled ventilation — After tracheal intubation, volume-controlled ventilation will be initiated with an I:E ratio of 1:2 and a tidal volume of 8 mL per ideal body weight (kg). Immediately after CO2 pneumoperitoneum with steep Trendelenburg positioning, Autoflow-volume controlled ventilation will be applied instead of volume-controlled ventilation. Immediately after CO2 desufflation and supine positioning, volume-controlled ventilation will be applied again.
  Other Names: Autoflow-VCV
  Arms: Autoflow-volume controlled ventilation

SUMMARY:
The steep trendelenburg position and pneumoperitoneum during laparoscopic surgery have the potential to cause an adverse effects on respiratory mechanics and gas exchange. Autoflow-volume controlled ventilation may improve lung compliance and reduce airway peak pressure. Therefore, the aim of this study is to evaluate whether Autoflow-volume controlled ventilation improves gas exchange and respiratory mechanics in patients undergoing robot-assisted laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients scheduled for elective robot-assisted laparoscopic radical prostatectomy undergoing general anesthesia

Exclusion Criteria:

1. chronic obstructive respiratory diseases
2. heart failure
3. body mass index (BMI >30 kg/m2)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
arterial oxygen tension (PaO2) | 30 minutes after steep trendelenburg position and pneumoperitoneum.
  Arterial oxygen tension (PaO2) obtained from arterial blood gas analysis

SECONDARY OUTCOMES:
The peak inspiratory pressure | 10 minutes after anesthesia induction, 30 and 60 minutes after steep trendelenburg position and pneumoperitoneum, and 10 minutes after supine position and CO2 desufflation.
  The peak inspiratory pressure during mechanical ventilation with endotracheal intubation under general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Background] Kim MS, Kim NY, Lee KY, Choi YD, Hong JH, Bai SJ. The impact of two different inspiratory to expiratory ratios (1:1 and 1:2) on respiratory mechanics and oxygenation during volume-controlled ventilation in robot-assisted laparoscopic radical prostatectomy: a randomized controlled trial. Can J Anaesth. 2015 Sep;62(9):979-87. doi: 10.1007/s12630-015-0383-2. Epub 2015 Apr 14. PMID 25869025